CLINICAL TRIAL: NCT00321984
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Dexlansoprazole MR (30 mg QD and 60 mg QD) Compared to Placebo on Symptom Relief in Subjects With Symptomatic Nonerosive Gastroesophageal Reflux Disease (GERD)
Brief Title: Safety and Efficacy of Dexlansoprazole Modified Release Formulation to Treat Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP Clinical Sciences, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-GD05-137; 2006-000420-13 (EudraCT Number); U1111-1114-1935 (Registry Identifier: WHO)
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2009-03-23 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease(GERD); Heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexlansoprazole MR 30 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Dexlansoprazole MR 60 mg QD (Experimental)
  Interventions: Drug: Dexlansoprazole MR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexlansoprazole MR — Dexlansoprazole MR 30 mg, capsules, orally, once daily for 4 weeks.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 30 mg QD
Drug: Dexlansoprazole MR — Dexlansoprazole MR 60 mg, capsules, orally, once daily for 4 weeks.
  Other Names: TAK-390MR; Kapidex; Dexilant
  Arms: Dexlansoprazole MR 60 mg QD
Drug: Placebo — Dexlansoprazole placebo-matching capsules, orally, once daily for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Dexlansoprazole modified release (MR) (30 mg once daily [QD] or 60 mg QD) compared to placebo in relief of daytime and nighttime heartburn over 4 weeks in subjects with symptomatic, nonerosive gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, multicenter, placebo-controlled, 3-arm study with a 4 week treatment period. This study will compare the efficacy of Dexlansoprazole MR (30 mg QD and 60 mg QD) with that of placebo when administered orally as a single daily dose in the morning, before breakfast. The study is designed to evaluate symptom relief in subjects with symptomatic nonerosive GERD. Approximately 900 subjects will be enrolled at approximately 200 United States (US) and potentially ex-US sites. The study consists of two periods: a screening period, which will last a minimum of 7 days and a maximum of 21 days, and a treatment period, which will last 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects identifying their main symptom as a burning feeling in the mid epigastric area and/or chest area (ie, heartburn).
* Subject has a history of episodes of heartburn for 6 months or longer prior to Screening.
* Subject must have a history of episodes of heartburn for 4 or more days during the 7 days prior to Day -1.

Exclusion Criteria:

* Endoscopic Barrett's esophagus and/or definite dysplastic changes. History of dilatation of esophageal strictures.
* Subjects with erosive esophagitis (EE) as shown by endoscopy.
* Evidence of uncontrolled systemic disease. Co-existing diseases affecting the esophagus. Current or history of Zollinger-Ellison syndrome.
* Subject has abnormal laboratory values.
* Subjects with active gastric or duodenal ulcers within 4 weeks of the first dose.
* Subject known to have acquired immunodeficiency syndrome (AIDS).
* Known hypersensitivity to any proton pump inhibitor (PPI), any component of Dexlansoprazole MR, or antacid.
* Use of prescription or non-prescription PPIs, histamine (H2) receptor antagonists, or sucralfate.
* Chronic (>12 doses per month) use of nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclo-oxygenase-2 (COX-2) inhibitors.
* Use of antacids (except for study-supplied Gelusil® ).
* Use of drugs with significant anticholinergic effects.
* Subjects who cannot discontinue the use of misoprostol or prokinetics
* Need for continuous anticoagulant therapy.
* Females who are pregnant or lactating.
* History of gastrointestinal surgery except for simple oversew of ulcer.
* History of cancer within 3 years prior to screening.
* Subject has participated in a previous Dexlansoprazole study.
* Subjects who, in the opinion of the investigator, are unable to comply with the requirements of the study or are unsuitable for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 947 (Actual)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (153):
- United States (153):
  - Alabaster, Alabama
  - Birmingham, Alabama
  - Hueytown, Alabama
  - Huntsville, Alabama
  - Northport, Alabama
  - Tallassee, Alabama
  - Chandler, Arizona
  - North Little Rock, Arizona
  - Sun City, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Azusa, California
  - Carmichael, California
  - Chula Vista, California
  - Clearwater, California
  - Cypress, California
  - Fountain Valley, California
  - Fullerton, California
  - Garden Grove, California
  - Irvine, California
  - Lancaster, California
  - Mission Hills, California
  - Oakland, California
  - Orange, California
  - Palm Springs, California
  - Pasadena, California
  - Redwood City, California
  - San Diego, California
  - San Francisco, California
  - San Luis Obispo, California
  - Vista, California
  - Westlake Village, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Littleton, Colorado
  - Lone Tree, Colorado
  - Wheat Ridge, Colorado
  - Bristol, Connecticut
  - Waterbury, Connecticut
  - Boynton Beach, Florida
  - Clearwater, Florida
  - Holly Hill, Florida
  - Jupitor, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Naples, Florida
  - New Smyma Beach, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Conyers, Georgia
  - Dunwoody, Georgia
  - Stockbridge, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Moline, Illinois
  - Oak Forrest, Illinois
  - Rockford, Illinois
  - Indianapolis, Indiana
  - Clive, Iowa
  - Dubuque, Iowa
  - Overland, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Hollywood, Maryland
  - Lutherville, Maryland
  - Prince Frederick, Maryland
  - Troy, Michigan
  - Chaska, Minnesota
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Jefferson City, Missouri
  - Mexico, Missouri
  - Washington, Missouri
  - Butte, Montana
  - Las Vegas, Nevada
  - Pahrump, Nevada
  - Egg Harbor Town, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Great Neck, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Harrisburg, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Franklin, Ohio
  - Kettering, Ohio
  - Lyndhurst, Ohio
  - Mogadore, Ohio
  - Sylvania, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Lansdale, Pennsylvania
  - Levittown, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Varnville, South Carolina
  - Sioux Falls, South Dakota
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Hermitage, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Beaumont, Texas
  - Bellaire, Texas
  - Bryan, Texas
  - Carollton, Texas
  - Conroe, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Midvale, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Norfold, Virginia
  - Richmond, Virginia
  - Lakewood, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin

REFERENCES:
- [Result] Fass R, Chey WD, Zakko SF, Andhivarothai N, Palmer RN, Perez MC, Atkinson SN. Clinical trial: the effects of the proton pump inhibitor dexlansoprazole MR on daytime and nighttime heartburn in patients with non-erosive reflux disease. Aliment Pharmacol Ther. 2009 Jun 15;29(12):1261-72. doi: 10.1111/j.1365-2036.2009.04013.x. Epub 2009 Apr 8. PMID 19392864
- [Result] Peura DA, Metz DC, Dabholkar AH, Paris MM, Yu P, Atkinson SN. Safety profile of dexlansoprazole MR, a proton pump inhibitor with a novel dual delayed release formulation: global clinical trial experience. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1010-21. doi: 10.1111/j.1365-2036.2009.04137.x. Epub 2009 Sep 4. PMID 19735233
- [Result] Friedlander EA, Pallentino J, Miller SK, VanBeuge SS. The evolution of proton pump inhibitors for the treatment of gastroesophageal reflux disease. J Am Acad Nurse Pract. 2010 Dec;22(12):674-83. doi: 10.1111/j.1745-7599.2010.00578.x. Epub 2010 Nov 24. PMID 21129076
- [Derived] Peura DA, Pilmer B, Hunt B, Mody R, Perez MC. Distinguishing the impact of dexlansoprazole on heartburn vs. regurgitation in patients with gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2013 Nov;38(10):1303-11. doi: 10.1111/apt.12504. Epub 2013 Sep 30. PMID 24118079
- [Derived] Peura DA, Pilmer B, Hunt B, Mody R, Perez MC. The effects of increasing body mass index on heartburn severity, frequency and response to treatment with dexlansoprazole or lansoprazole. Aliment Pharmacol Ther. 2013 Apr;37(8):810-8. doi: 10.1111/apt.12270. Epub 2013 Mar 4. PMID 23451835
- See also: For the Dexilant package insert refer to this link — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled at 154 sites in the United States (US); date of first dose: 08 June 2006; date of last procedure: 11 December 2006.
Pre-assignment Details: Subjects with endoscopically documented normal esophageal mucosa were enrolled in Dexlansoprazole Modified Release (MR) or Placebo once daily (QD) treatment group; subjects were instructed that lifestyle or behavioral modifications designed to treat their symptoms of gastroesophageal reflux disease (GERD) should not be altered throughout the study.
Groups:
- Placebo QD: Placebo capsules, orally, once daily for up to 4 weeks.
- Dexlansoprazole MR 30 mg QD: Dexlansoprazole MR 30 mg, capsules, orally, once daily for up to 4 weeks.
- Dexlansoprazole MR 60 mg QD: Dexlansoprazole MR 60 mg, capsules, orally, once daily for up to 4 weeks.
Period: Overall Study
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Started | 317 | 315 | 315
Completed | 290 | 294 | 289
Not Completed | 27 | 21 | 26
Not completed — Adverse Event | 9 | 6 | 8
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 4 | 2
Not completed — Withdrawal by Subject | 8 | 6 | 5
Not completed — Unmet Inclusion/Exclusion Criteria | 3 | 1 | 5
Not completed — Lack of Efficacy | 3 | 1 | 3
Not completed — Noncompliant | 0 | 0 | 2
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Per Subject Request | 1 | 0 | 0
Not completed — Per Investigator Request | 1 | 0 | 0
Not completed — Per Sponsor Due to High Baseline Gastrin | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD | Total
Number analyzed (Participants) | 317 | 315 | 315 | 947
Age Continuous [Mean (Standard Deviation); unit: years] | 47.6 (14.40) | 47.6 (13.55) | 47.5 (13.77) | 47.5 (13.90)
Age, Customized [Number; unit: participants]
  <45 years | 130 | 131 | 139 | 400
  45 to <65 years | 148 | 149 | 136 | 433
  ≥65 years | 39 | 35 | 40 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 231 | 209 | 673
  Male | 84 | 84 | 106 | 274
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 2 | 5
  Asian | 5 | 4 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 0 | 4
  Black or African American | 45 | 37 | 48 | 130
  White | 255 | 267 | 251 | 773
  More than one race | 4 | 3 | 6 | 13
  Unknown or Not Reported | 2 | 3 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 67 | 53 | 182
  Not Hispanic or Latino | 255 | 248 | 262 | 765
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days With Neither Daytime Nor Nighttime Heartburn During Treatment as Assessed by Daily Electronic Diary-Median
Description: The percentage was calculated as the days that were heartburn-free out of the total number of days for which either a daytime or nighttime result was marked.
Time Frame: 4 weeks
Population: Analysis was conducted on an intent-to-treat (ITT) population that included all randomized subjects who received at least 1 dose of study drug and completed at least 1 diary entry for heartburn during treatment. All ITT populations excluded subjects with confirmed Barrett's esophagus and/or definite dysplastic changes.
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 310 | 312 | 307
percentage of days | 18.5 [0.0 to 42.9] | 54.9 [19.7 to 80.9] | 50.0 [14.8 to 80.6]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 30 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — The overall 0.0025 level of significance for the multiple comparisons of each dexlansoprazole MR dose to placebo was controlled using Hochberg's method
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.72941, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.0025 level without adjustment for multiple comparisons

2. Primary Outcome: Percentage of Days With Neither Daytime Nor Nighttime Heartburn During Treatment as Assessed by Daily Electronic Diary-Mean
Description: as for outcome 1
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 310 | 312 | 307
percentage of days | 25.0 (25.6) | 50.3 (33.9) | 49.1 (34.7)

3. Secondary Outcome: Percentage of Days Without Nighttime Heartburn During Treatment as Assessed by Daily Electronic Diary-Median
Description: The percentage was calculated as the nights that were heartburn-free out of the total number of days for which a nighttime result was marked.
Time Frame: 4 weeks
Population: Analysis was conducted on an ITT population (all randomized subjects who received at least 1 dose of study drug and completed at least 1 diary entry for heartburn during treatment), but excluded subjects without any morning diary entries on Day 1 or later.
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 308 | 311 | 307
percentage of days | 51.7 [16.3 to 74.3] | 80.8 [45.8 to 95.8] | 76.9 [43.3 to 94.4]
Statistical Analysis 1: Comparison: Placebo QD vs Dexlansoprazole MR 30 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Dexlansoprazole MR 60 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dexlansoprazole MR 30 mg QD vs Dexlansoprazole MR 60 mg QD; The comparison between the two treatment groups was made using Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.31460, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.0025 level without adjustment for multiple comparisons

4. Secondary Outcome: Percentage of Days Without Nighttime Heartburn During Treatment as Assessed by Daily Electronic Diary-Mean
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Number analyzed (Participants) | 308 | 311 | 307
percentage of days | 47.1 (32.6) | 67.6 (34.1) | 65.0 (34.3)

ADVERSE EVENTS:
Arm/Group | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Serious Adverse Events (participants affected / at risk) | 1 | 2 | 1
Other Adverse Events (participants affected / at risk) | 34 | 41 | 36
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Coronary Artery Disorders Not Elsewhere Classified (NEC) (Cardiac disorders) | 1/317 | 0/315 | 0/315
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 0/317 | 2/315 | 0/315
Heart Failures NEC (Cardiac disorders) | 0/317 | 1/315 | 0/315
Sepsis, Bacteraemia, Viraemia and Fungaemia NEC (Infections and infestations) | 0/317 | 1/315 | 0/315
Gastrointestinal & Abdominal Pains (Excluding Oral and Throat) (Gastrointestinal disorders) | 0/317 | 0/315 | 1/315
Non-site Specific Gastrointestinal Haemorrhages (Gastrointestinal disorders) | 0/317 | 0/315 | 1/315
Central Nervous System Haemorrhage & Cerebrovascular Accidents (Nervous system disorders) | 0/317 | 1/315 | 0/315
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo QD | Dexlansoprazole MR 30 mg QD | Dexlansoprazole MR 60 mg QD
Diarrhoea (Excluding Infective) (Gastrointestinal disorders) | 11/317 | 18/315 | 15/315
Headaches NEC (Nervous system disorders) | 19/317 | 13/315 | 9/315
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 9/317 | 16/315 | 18/315

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.